CLINICAL TRIAL: NCT03156179
Title: Assessment of Calcium Metabolism in Adolescent Girls With Type 1 Diabetes
Brief Title: Study of Calcium Metabolism in Teenage Girls With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Cornell University (Other)
Responsible Party: Principal Investigator, David Weber, Assistant Professor, University of Rochester
Other Study IDs: 56744
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Girls with type 1 diabetes
  Interventions: Diagnostic Test: calcium isotope analysis

INTERVENTIONS:
Diagnostic Test: calcium isotope analysis — A dual stable calcium isotope method will be used to determine fractional calcium absorption. Two stable calcium isotopes will be administered to participants in order to determine fractional calcium absorption. 7 mg of 44Ca will be administered orally in 60 mL of liquid at the start of the study. 2 mg of 42Ca will then be administered intravenously. 24 hour urine collection will begin immediately following oral tracer administration for the assessment of urinary calcium excretion. The enrichment of 44Ca and 42Ca in urine will be determined by magnetic sector thermal ionization mass spectrometry. The isotopic ratios of 44Ca and 42Ca to 48Ca (another naturally occurring calcium isotope present in the human body) will be calculated (42Ca/48Ca and 44Ca/48Ca). The relative fraction of the oral to intravenously administered isotope in the 24 hour urine sample [(42Ca/48Ca) / (44Ca/48Ca)] is the fractional calcium absorption.

SUMMARY:
The proposed pilot study will enroll 33 adolescent females with type 1 diabetes for the assessment of whole body calcium metabolism using dual stable calcium isotopes. This is the state of the art technique for assessing calcium metabolism in the body and has been used in both healthy and diseased pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D of at least three years duration
* Female sex
* Age between 9-18 years
* Parental/guardian consent and participant assent
* BMI <99th percentile

Exclusion Criteria:

* History of metabolic bone disease, chronic renal disease, hepatic disease, celiac, or other malabsorptive disease
* History of any proton-pump inhibitor use within a 6 month period prior to enrollment
* History of oral or inhaled corticosteroid use for ≥ 5 consecutive days within a 6 month period prior to enrollment
* Pregnant or lactating females
* Parents/guardians or participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 9 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Females has an increased risk of bone fractures.
Study Population: Teenage girls with type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
fractional calcium absorption | 24 hours
  Mass spectroscopy was performed using urine to measure the stable calcium isotope. Percent dietary calcium absorption was calculated as the ratio of the cumulative recovery of 44Ca (oral tracer) to the cumulative recovery of 42Ca (IV tracer) in the 24-hour urine sample.

SECONDARY OUTCOMES:
Estimated calcium retention | 24 hours
  Gastrointestinal calcium absorption minus the total of urine calcium excretion and estimated stool calcium excretion.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weber DR, O'Brien KO, Schwartz GJ. Evidence of disordered calcium metabolism in adolescent girls with type 1 diabetes: An observational study using a dual-stable calcium isotope technique. Bone. 2017 Dec;105:184-190. doi: 10.1016/j.bone.2017.09.001. Epub 2017 Sep 4. PMID 28882565